CLINICAL TRIAL: NCT03545685
Title: Enhancing Intervention of Attenuated Psychosis Syndrome With M-Health Technology
Brief Title: Intervention of Attenuated Psychosis Syndrome With M-Health Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida A&M University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 005680
Record Dates: First submitted 2018-05-04; First posted 2018-06-04 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-07

CONDITIONS: Adolescent - Emotional Problem

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SMART (Experimental): The subjects in SMART training group will receive add-on SMART intervention for 3 months. Subjects will play cognitive games for 1 hour per day, five days per week. SMART will track game time, resource use, and text messaging information on a daily basis, which allows researchers/clinicians to monitor subjects' daily SMART activities. Daily end-of-day RedPocket incentives will be delivered to subjects' designated account based on their resource use and game time. Top 5 APS subjects who play the game for the most time in a week will be rewarded
  Interventions: Other: specific memory and attention realtime training
- Control group (Other): Participants in this group will serve as control group
  Interventions: Other: specific memory and attention realtime training

INTERVENTIONS:
Other: specific memory and attention realtime training — The investigator will conduct a pilot study of 80 APS subjects (age 18-45). The investigator will examine SMART feasibility and user engagement using a randomized control trial research design. Using a simple random method, 40 APS subjects will be randomly assigned to the experimental group to receive add-on SMART intervention for 3 months and 40 APS subjects will just get naturalistic treatment with no SMART intervention. At baseline and 3-month follow-up, subjects will complete questionnaires on app use habits and attitudes towards SMART feasibility and engagement. In-depth interviews will be conducted at both time points to cross-validate the findings obtained from the questionnaires.

SUMMARY:
The investigators will develop a culturally sensitive smart phone application to enhance neurocognitive function (memory and attention in particular) of participants with attenuated psychosis syndrome (APS).

DETAILED DESCRIPTION:
The investigator will conduct a pilot study of 80 APS subjects (age 18-45). Forty subjects will be randomly put in the SMART plus routine care (RC) group and 40 to RC group only. At baseline and 3-month follow-ups, all subjects will complete questionnaires including Mobile App Rating Scale SMART feasibility and engagement. 1:1 in-depth interviews will be conducted at the two time points to cross-validate the findings obtained from the questionnaires. The questionnaires and in-depth interviews for APS subjects for the RC group seek to explore their preference and likelihood to use SMART given the opportunity. Examine Cognitive Function Change. In order to prepare for future large scale randomized clinical trials, the investigator will examine the effectiveness of SMART in improving working memory and attention of APS subjects. At baseline and 3-month follow-ups, all subjects will complete MATRICS Consensus Cognitive Battery (MCCB) subtests measuring working memory (Spatial Span) and attention (Continuous Performance Test-Identical Pairs). A between and within group design allows examining change of outcome variables over time and group differences. Enhance mHealth research capacity of SMHC at individual and organization levels.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 45 years old.
* Understand and sign an informed consent (or assent for minors) document.
* Must meet the substance use criteria: No DSM IV Alcohol or Drug Dependence in the past 3 months; No use on the day of assessment, clearly not high or hung-over.
* Meet diagnostic criteria for a prodromal syndrome. If under the age of 19 and meets diagnostic criteria for Schizotypal Personality Disorder or meets the diagnostic criteria called the Criteria for Prodromal Syndromes (COPS) which are operationalized as follows:

  * Genetic Risk and Deterioration Syndrome (GRDS): First degree relative with psychosis or subject with Schizotypal Personality Disorder and a 30% drop in GAF score compared to one year ago, sustained over the past month, or
  * Attenuated Positive Symptoms Syndrome (APSS): Severity rating of moderate (rating of 3), moderately severe (4) or severe but not psychotic (5) on any one of the five SOPS positive symptoms; symptom occurs at above severity level at an average frequency of at least once per week in the past month; symptom must have begun in the past year or currently rates at least one scale point higher than rated 12 months previously, or
  * Brief Intermittent Psychotic Syndrome (BIPS): Severity rating of psychotic intensity (6) on any of the 5 SOPS positive symptoms 94; symptom is present at least several minutes per day at a frequency of at least once per month; symptom(s) must have reached a psychotic intensity in the past 3 months; symptom is not seriously disorganizing or dangerous; symptom(s) do not last for more than 1 hour/day at an average frequency of 4 days/week over 1 month.

Exclusion Criteria:

* Meet criteria for current or lifetime Axis I psychotic disorder, including affective psychoses and psychosis NOS.
* Impaired intellectual functioning (i.e. IQ<70).
* Past or current history of a clinically significant central nervous system disorder that may contribute to prodromal symptoms or confound their assessment.
* Traumatic Brain Injury that is rated as 7 or above on the Traumatic Brain Injury screening instrument (signifying a significant brain injury with persistent sequelae).
* The diagnostic prodromal symptoms are clearly caused by an Axis 1 disorder, including substance use disorders, in the judgment of the evaluating clinician. Other non-psychotic disorders will not be exclusionary (e.g. substance abuse disorder, major depression, anxiety disorders, Axis II Disorders), as long as the disorder does not account for the diagnosis of prodromal symptoms.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Memory and attention scores | 3rd month
  Memory and attention score will be assessed at 3 month followup

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mental Health Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided